CLINICAL TRIAL: NCT07273396
Title: A Phase 1/2a Study to Evaluate the Tolerance, Safety, Efficacy, and Pharmacokinetics of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Using Paclitaxel for Platinum-resistant Recurrent Ovarian Cancer With Peritoneal Metastasis (PIPAC-OVPAC 1/2a)
Brief Title: Tolerance, Safety, Efficacy, and Pharmacokinetics of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Using Paclitaxel for Platinum-resistant Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC-OVPAC-1/2a
Record Dates: First submitted 2025-05-05; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms
Keywords: Pressurized intraperitoneal aerosol chemotherapy; platinum-resistant recurrent; ovarian cancer; paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIPAC-OVPAC group (Experimental)
  Interventions: Drug: Pressurized intraperitoneal aerosol chemotherapy (PIPAC) using paclitaxel

INTERVENTIONS:
Drug: Pressurized intraperitoneal aerosol chemotherapy (PIPAC) using paclitaxel — All patients enrolled in this study receive PIPAC using paclitaxel under 12 mmHg at 6 weeks intervals (up to 9 cycles)
  1. Phase 1 Design
     1. Dose Escalation: Standard 3+3 design across 5 paclitaxel cohorts (20 → 40 → 67 → 100 → 140 mg/m²) using modified Fibonacci increments (100%, 67%, 50%, 40%).
     2. Maximum tolerated dose(MTD) Determination
        * If ≥2/6 patients in cohort χ experience dose limiting toxicities(DLTs; Grade ≥3 toxicity per CTCAE v5.0, excluding manageable pain) and ≤1/6 in cohort χ-1, MTD = χ-1.
        * If no DLTs at 140 mg/m², Phase 1 concludes.
     3. Dose Reduction
        * DLTs in 20 mg/m² trigger de-escalation to 10 mg/m².
        * If ≤1/6 DLTs in 10 mg/m² → RP2D; ≥2/6 DLTs → trial termination.
  2. Phase 2 Design : Evaluates efficacy/safety of PIPAC at the RP2D in 23 patients, adjusting for 5-17% laparoscopic access failure.

SUMMARY:
The purpose of this study is to evaluate the tolerance, safety, efficacy, and pharmacokinetics of pressurized intraperitoneal aerosol chemotherapy (PIPAC) with paclitaxel in patients with platinum-resistant recurrent ovarian cancer and peritoneal carcinomatosis.

DETAILED DESCRIPTION:
The Study Design is an interventional, non-randomized, sequential Phase 1/2a trial, where patients with platinum-resistant recurrent ovarian cancer(PROC) and radiologically confirmed peritoneal carcinomatosis will be enrolled.

All patients included in this study will receive PIPAC, laparoscopic aerosolization of paclitaxel under 12 mmHg pressure at 6-week intervals (up to 9 cycles) for treating PROC with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Women aged 19-85 years.
2. Diagnosis: Histologically confirmed ovarian, fallopian tube, or peritoneal cancer.
3. Platinum Status:

   * Refractory: Disease progression during platinum-based chemotherapy.
   * Resistant: Progression within 6 months (24 weeks) post-platinum therapy.
4. Prior Therapies: ≥2 prior intravenous chemotherapies (may include paclitaxel).
5. Treatment Options: Unresponsive to/ineligible for standard therapies (e.g., intolerance, hypersensitivity) and ineligible for surgical resection.
6. Measurable Disease: ≥1 measurable/evaluable peritoneal lesion per RECIST 1.1.
7. Metastasis: ≤1 asymptomatic distant metastasis (excluding retroperitoneal lymph nodes, pleural effusion, localized skin metastases).
8. Imaging Confirmation: Peritoneal carcinomatosis confirmed by PET-CT/CT.
9. Performance Status: ECOG 0-2.
10. Pregnancy/Contraception:

    * Non-pregnant/non-lactating.
    * Contraception: Effective methods (IUD, sterilization) for 6 months post-PIPAC (childbearing potential only).
11. Organ Function:

    * Bone Marrow: ANC >1,500/mm³, platelets >100,000/mm³, hemoglobin >8.0 g/dL.
    * Liver: Bilirubin ≤1.5×ULN, AST/ALT ≤1.5×ULN.
    * Kidney: Creatinine ≤1.5×ULN, creatinine clearance >60 mL/min.
    * Lungs: FVC/FEV1 ≥70% predicted.
    * Coagulation: INR ≤1.5, aPTT ≤1.5×ULN.
12. Consent: Signed informed consent.

Exclusion Criteria:

1. ≥2 distant metastases (excluding retroperitoneal lymph nodes, pleural effusion, and localized skin metastases).
2. Contraindications to paclitaxel per approved domestic labeling.
3. Hypersensitivity history to paclitaxel or PIPAC devices.
4. Uncontrolled comorbidities per investigator judgment:

   * NYHA Class ≥II heart failure
   * Clinically significant cardiovascular disease (e.g., arrhythmia, myocardial infarction)
   * Immunosuppressive conditions (AIDS, autoimmune diseases, immunosuppressive therapy)
   * Active HBV/HCV infection
   * Uncontrolled hypertension (systolic >160 mmHg or diastolic >100 mmHg)
   * Uncontrolled diabetes (HbA1c >8%)
   * Radiographic/clinical bowel obstruction.
5. IV chemotherapy within 4 weeks prior to Cycle 1 PIPAC.
6. Life expectancy <3 months.
7. Prior PIPAC therapy.
8. Medically unfit for general anesthesia or laparoscopic surgery.
9. Refusal of contraception:

   - Medically acceptable methods:
   * Intrauterine device (failure rate <1%)
   * Surgical sterilization (tubal ligation, hysterectomy, vasectomy; failure rate <0.5%).
10. Participation in another clinical trial within 1 month of screening.
11. Other exclusionary factors per investigator discretion.

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities | Till 6 weeks after the first PIPAC in phase 1 study
  Dose limiting toxicities
Maximum tolerated dose | During phase 1 study (up to 6 weeks)
  We consider dose escalation if 3 consecutive DLTs do not occur, or less than 1 in 6 DLTs occur, per standard 3+3 design. If DLT occurs in 2 or more of 6, the lower dose is considered the MTD if 1 or fewer DLTs are identified. In addition, the highest dose (140 mg/m2) is considered the MTD when 3 to 0 DLTs or 6 to 1 DLTs are identified at the highest dose. On the other hand, if the initial dose (20 mg/m2) is reduced to 10 mg/m2 to account for DLT, it is considered the MTD if no more than 1 in 6 develop DLT at that reduced dose.
Recommended Phase 2 Dose | During phase 1 study
  Recommended Phase 2 Dose determined by dose limiting toxicities
Disease control rate | During phase 2 study
  Disease control rate at the 9-week time point

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | During phase 1 study
  Cmax on pharmacokinetic evaluation of paclitaxel administered via pressurized intraperitoneal aerosol chemotherapy
Time at which Cmax is observed (Tmax) | During phase 1 study
  Tmax on pharmacokinetic evaluation of paclitaxel administered via pressurized intraperitoneal aerosol chemotherapy
Area under the curve (AUC) | During phase 1 study
  AUC on pharmacokinetic evaluation of paclitaxel administered via pressurized intraperitoneal aerosol chemotherapy
Disease control rate | During phase 1 study
  Disease control rate at the 9-week time point
Progression-free survival | During phase 1 and 2a studies
  Time from the treatment start of pressurized intraperitoneal aerosol chemotherapy to the identification of progressive disease or the end of the study
Overall survival | During phase 1 and 2a studies
  Time from the treatment start of pressurized intraperitoneal aerosol chemotherapy to cancer-related death or the end of the study
Peritoneal cancer index | During phase 1 and 2a studies
  Peritoneal cancer index scores identified during pressurized intraperitoneal aerosol chemotherapy, which range from 0 to 39
Peritoneal Regression Grading Score | During phase 1 and 2a studies
  Peritoneal Regression Grading Score examined by pathologic review; Peritoneal Regression Grading Score 1, complete response: Peritoneal Regression Grading Score 2, major response: Peritoneal Regression Grading Score 3, minor response; Peritoneal Regression Grading Score 4, no response
Changes in ascites volume | During phase 1 and 2a studies
  Changes in ascites volume measured during pressurized intraperitoneal aerosol chemotherapy
CA-125 | Assessed at every visit during the study period
  Seum CA-125 levels, which are related to disease progression when more than 35 U/ml
human epididymis protein 4 (HE4) | Assessed at every visit during the study period
  Serum HE4 levels, which are related to disease progression when more than 140 pmol/L
The Risk of Ovarian Malignancy Algorithm (ROMA) score | Assessed at every visit during the study period
  ROMA score using serum CA-125 and HE4 levels, which are related to disease progression when more than 30%
EORTC QLQ-C30 questionnaire | During phase 1 and 2a studies
  EORTC QLQ-C30 questionnaires measured during the study. The evaluation range for each item is from 0 to 100.
EORTC QLQ-OV28 questionnaire measured during the study | During phase 1 and 2a studies
  EORTC QLQ-OV28 questionnaire measured during the study. The evaluation range for each item is from 0 to 100.
Safety evaluation | During phase 1 and 2a studies
  Safety evaluation per CTCAE v5.0, including treatment-related adverse events and surgical complications. The evaluation range for each item is from grade 1 to grade 5.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD, PhD, Principal Investigator — Seoul National University College of Medicine

IPD SHARING:
Plan to Share IPD: No